CLINICAL TRIAL: NCT07240259
Title: Feasibility of Tracheobronchial Reconstruction Using Allogenic Aortic Patch in Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202404094DINC
Record Dates: First submitted 2025-09-12; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Trachea Diseases; Tracheal Stenosis; Tuberculosis; Tracheitis; Airway Disease; Tracheomalacia; Tracheal Stenosis Following Tracheostomy; Tracheal Reconstruction Surgery
Keywords: tracheomalacia; bronchial reconstruction; cryopreserved aorta; tracheal reconstruction; tracheal stenosis
MeSH Terms: conditions — Tracheal Diseases; Tracheal Stenosis; Tuberculosis; Tracheitis; Tracheomalacia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryopreserved aorta (Experimental): After resection of tracheal or bronchial lesion, reconstruct the airway with cryopreserved aortic allograft.
  Interventions: Procedure: Cryopreserved aorta

INTERVENTIONS:
Procedure: Cryopreserved aorta — After resection of the tracheal or bronchial lesion with standard surgical techniques, the airway gap is reconstructed with a segment of human cryopreserved (-80 celsius degree) aortic allograft, which was not matched by the ABO and leukocyte antigen systems. The anastomosis is performed with standard technique for airway anastomosis.

SUMMARY:
Feasibility and safety of repairing tracheal and bronchial defects in infants and children using cryopreserved donor aortic patches.

DETAILED DESCRIPTION:
This trial plans to use cryopreserved donor aortic tissue patches to repair and treat pediatric patients with end-stage, life-threatening or severely disabling tracheal diseases who have not responded to conventional conservative therapies or lack sufficient native tracheal tissue for tracheal defect reconstruction.

ELIGIBILITY:
Inclusion Criteria:

Meeting any of the following conditions, and being unsuitable for standard end-to-end tracheal anastomosis or lacking sufficient native tracheal tissue for defect reconstruction:

1. Congenital tracheal malformations: including congenital tracheomalacia, congenital tracheobronchial anomalies, complete tracheal rings, etc., with severe clinical respiratory symptoms and recommended for treatment after evaluation.
2. Acquired tracheal stenosis: including tracheal narrowing caused by disease, endotracheal intubation, or postoperative scar formation, with severe clinical respiratory symptoms and recommended for treatment after evaluation.
3. Tracheal injury or tissue loss due to trauma or burns requiring surgical repair.
4. Tracheal tumors: reconstruction of tracheal tissue after resection of benign or malignant tumors.
5. The term "severe clinical respiratory symptoms" includes:

   1. Dependence on mechanical ventilation for more than 1 month due to airway narrowing or defect, with inability to wean.
   2. Airway stenosis exceeding 50% (confirmed by bronchoscopy or CT imaging), accompanied by persistent stridor, inspiratory dyspnea, or suprasternal/substernal retractions, causing impairment of daily activities or feeding difficulties.
   3. Unilateral or bilateral lung atelectasis persisting for more than 1 month due to tracheal or bronchial stenosis, with no sign of recovery.
   4. Recurrent post-obstructive pneumonia (≥3 episodes) in one or both lungs caused by tracheal or bronchial stenosis, requiring hospitalization for treatment.

Exclusion Criteria:

1. Inability to obtain legal informed consent from the lawful guardian.
2. Locally invasive tracheal tumors that cannot be completely resected surgically.
3. Malignant solid tumors with distant metastases that cannot be completely resected surgically or controlled with medication.
4. Presence of severe immunodeficiency (e.g., congenital immunodeficiency, HIV infection, ongoing chemotherapy, or recovery period after bone marrow transplantation).
5. Presence of major congenital diseases or chromosomal abnormalities (e.g., Trisomy 13, Trisomy 18) with extremely poor prognosis as assessed clinically.
6. End-stage organ failure (e.g., persistent multiple organ failure, irreversible cardiopulmonary failure, or brain death).

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
90-day Mortality | Postoperative 90 days
  Survival status of patients within 90 days after surgery. This primary endpoint evaluates patient mortality, as patients undergoing this type of surgery often have a high short-term risk of death.

SECONDARY OUTCOMES:
Anastomotic Leakage | Within 90 days postoperatively
  Incidence of anastomotic leakage at the tracheal anastomosis site.
Pneumonia | Within 90 days postoperatively
  Incidence of postoperative pneumonia.
Difficult Extubation | Within 90 days postoperatively
  Occurrence of difficulties in extubation after surgery.
Granulation Tissue Obstruction | Within 90 days postoperatively
  Incidence of airway obstruction due to granulation tissue formation.
Stenosis Caused by Scar Fibrosis and Related Complications | Within 90 days postoperatively
  Occurrence of airway stenosis due to scar fibrosis or other related complications.

OTHER OUTCOMES:
Long-term Clinical Follow-up | At least 1 year postoperatively; infants and young children followed until at least puberty
  Patients will undergo long-term follow-up including medical history review, physical examination, and imaging studies as clinically indicated (including but not limited to X-ray, CT scan, and bronchoscopy) to monitor long-term airway status and overall health.

CONTACTS AND LOCATIONS:
Locations (1):
- Taiwan National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsou KC, Hung WT, Ju YT, Liao HC, Hsu HH, Chen JS. Application of aortic allograft in trachea transplantation. J Formos Med Assoc. 2023 Sep;122(9):940-946. doi: 10.1016/j.jfma.2023.03.006. Epub 2023 Mar 29. PMID 37002174
- [Background] Lu CW, Liao HC, Tsou KC, Hung WT, Huang PM, Hsu HH, Chen JS. Cryopreserved aortic graft patch repair of traumatic tracheal rupture defect: A case report. JTCVS Tech. 2024 Aug 17;27:182-184. doi: 10.1016/j.xjtc.2024.07.023. eCollection 2024 Oct. No abstract available. PMID 39478918
- [Background] Hung WT, Liao HC, Hsu HH, Chen JS. Stented cryopreserved aortic allograft for reconstruction of long-segment post-tuberculosis tracheal stenosis. J Formos Med Assoc. 2024 Jul;123(7):818-820. doi: 10.1016/j.jfma.2024.03.006. Epub 2024 Mar 16. PMID 38494361